CLINICAL TRIAL: NCT00172926
Title: Cross Sectional Study on Relationship Between Physical Constitution and Diseases in the Integrative Chinese Medicine and Western Medicine
Brief Title: Study on the Relationship Between Physical Constitution and Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700326
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-12-21 (Estimated); Status verified 2005-06

CONDITIONS: Chronic Diseases
Keywords: Physical Constitution; Disease Pattern; Laboratory Data; Integrative Chinese Medicine and Western Medicine
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Physical constitution is an important factor for the development and outcome of diseases according to the theory in traditional Chinese medicine.

The purpose of the study is to find the correlation between physical constitution and clinical characteristics (age, sex, symptoms, physical signs, life style, laboratory results and image findings) through the questionnaire and results of health examination.

DETAILED DESCRIPTION:
It is difficult to predict the process or outcome of disease for individuals who expose to the same pathogen or condition. But according to the Traditional Chinese Medicine, physical constitution is an important factor for disease pattern, severity and response to the treatment. So it is paid more and more attention in Western Medicine to study the variation of individualized susceptibility to diseases.

There have been some researches to investigate the relationship between physical constitution and disease pattern. Before further studies, we need to obtain more information about physical constitution and clinical characteristics. Therefore we design a comprehensive questionnaire to survey the types of physical constitution. And we plan to collect the data from health reports of candidates after their medical tests at Health Examination Center in National Taiwan University Hospital Yu-Lin Branch. We focus on the relationship between clinical characteristics (age, sex, symptoms, physical signs, laboratory results and image findings) of Western Medicine and the physical constitutional types of Chinese Medicine. Then we will try to find the correlation and significance between them.

The study will conclude the constitutional characteristics in general population of Taiwan and the distribution tendency of physical constitution for the common diseases. The result can serve as a stepping stone for integration of the Traditional Chinese Medicine and Western Medicine.

ELIGIBILITY:
Inclusion Criteria:

* candidates with healthy report on health exam

Exclusion Criteria:

* acute infection
* chronic disease with acute exacerbation
* unstable disease status or medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2005-05; Study Completion 2007-04

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chang Su, PhD, Study Director — China Medical University, China
Locations (1):
- National Taiwan University Hospital Yun-Lin Branch, Douliu, Taiwan